CLINICAL TRIAL: NCT05316285
Title: Effects of School-based Yoga Program on University Students on Physical, Emotional and Psychosocial Health
Brief Title: Effects of School-based Yoga Program on University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Pınar KAYA, Assistant Professor, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-1950
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Yoga; Adolescent Behavior; Emotional Regulation; Mental Health; Eating Behaviors; Well-being
MeSH Terms: conditions — Adolescent Behavior; Emotional Regulation; Psychological Well-Being; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): It will consist of students who choose the Yoga for a Healthy Life lesson. For 14 weeks, one day a week and 60 minutes a day, theoretical and practical yoga training will be applied.
  Interventions: Other: Yoga exercise
- Control Group (No Intervention): The control group will consist of students who chose the Fashion and Beauty lesson.

INTERVENTIONS:
Other: Yoga exercise — Yoga lesson practices will be designed and implemented by instructors physiotherapists who have completed 200 hours of yoga instructor training (RYT-200). The yoga program, which will consist of one-hour sessions once a week, is planned to last 14 weeks. 4 weeks of classes will be theoretical lessons related to yoga philosophy, 10 weeks of yoga sessions will be applied every week on different concepts such as upper extremity and / or lower extremity focused strengthening and / or flexibility and breathing exercises. In addition to this training, students will be advised to repeat the practices once a week. Sessions will begin with breathing practices called pranayama, followed by yoga postures called asanas, and the sequence will be finished with savasana pose. In this pose, guided meditations will be performed on subjects such as body awareness and self-compassion.
  Arms: Yoga Group

SUMMARY:
Focusing on emotions is valuable because "how a person feels, reacts, and expresses emotions can have both short-term and long-term effects on physical and mental health". This is explained by mechanisms such as reappraisal, attention regulation, self-monitoring, self-awareness, and regulation of the autonomic nervous system. Because yoga reduces negative emotions such as anxiety, anger, and depression, teens are likely to result in less conflict and stress in their lives. It is thought that it is also important for young people to accept difficult feelings and to be able to accept and approve these feelings. When negative emotions are acknowledged and witnessed, they often dissolve or transform, and the process allows the individual to learn about their limits, preferences, and needs. Processing emotions in this way allows a person to be honest with oneself and can contribute to healthier development. Therefore, yoga appears to be a useful well-being tool and practice that schools should adopt, as it can increase life skills for students such as concentration, memory, relational skills, and decision-making that are affected by emotions. Emotional well-being is important for learning in life and school. As noted earlier, research supports such a view, but more research is needed to understand how and why yoga should be offered to young people in their schools. However, it is suggested that researchers further explore the role of yoga in the management of emotions, both in terms of emotional processing and regulation of emotions. The role of yogic breathing (pranayama) as part of a holistic perspective on yoga, and specifically the role of yoga in the relationship between being with emotions, regulating emotions, and how it relates to change, should be further explored.

It has been described in the literature that care should be taken to avoid possible harm to individuals associated with the use of unhealthy weight control behaviors among young adults and women with obesity. Yoga's intent to strengthen and support a positive sense of self makes it a particularly viable strategy for healthy weight management for women and those at high risk for poor body image. Finally, it has been reported that reductions in perceived stress may mediate the effects of participation in a yoga program on negative emotional and behavioral problems. It has been suggested that future studies may also assess the extent to which exposure to stress and trauma may affect youth's participation in and benefit from mindfulness and yoga interventions.

Considering all the suggestions and research needs in the literature, this study was planned to examine the improvement in self-esteem, life satisfaction, body image, anxiety, depression and cognitive emotion regulation levels of university students after their participation in the yoga program provided to them in the school environment and to compare them with students who do not do yoga. In the study, it is planned to investigate the pre-exam anxiety levels of university youth who regularly practice yoga.

DETAILED DESCRIPTION:
Adolescence is often described as a period of hypersensitivity that includes increased risk-taking and reward seeking. Such a period of high emotionality will often affect the well-being and mental health of young people, as some experiences can be like emotional roller coasters. Adolescence is not only a period of increased emotionality, but also a psychopathology related to affect. Therefore, how teens relate to their emotions is important to their overall well-being. Young individuals face many internal and external changes that can make them overly emotional. In general, the teenage years are characterized by emotional turmoil, as there is more activation in the emotional part of the brain (limbic system) during adolescence. It has been reported that adolescents are highly emotional, therefore they are often "captured by their emotions" and that the emotional life of adolescents is quite complex both internally and externally. On the inside, teens experience both hormonal changes and "fine-tuning of the neural networks that both generate and govern their emotions". From the outside, young people often experience dramatic changes in their social relationships (parents, peers, romantic relationships, etc.) with the increasing demands of school and society. Because of this high level of emotionality, the adolescence years are characterized by "increased psychopathological levels of dysfunctional affect". Learning to manage emotional responses is an important developmental task for young people's socio-cognitive development. Their development in these areas will affect their emotional decision-making and self-regulation skills.

Miller et al. in their review confirm that yoga is a promising intervention for children and youth. Researchers have also reported that "yoga has positive effects on a range of outcomes in psychological/behavioral, cognitive, and physiological/physical functioning." Researchers have reported that practicing yoga can improve mental health and well-being in school settings and beyond, and that yoga facilitates learning among young people. While schools are highlighted as ideal environments for promoting healthy lifestyle skills from an early age, there is less clarity about yoga styles, advice on frequency, and how it works. Still, scholars seem to agree on the value of teaching yoga as a holistic system of practice, including asanas or physical postures, pranayama or breathing exercises, relaxation techniques, and meditation or mindfulness practices.

Young people's mental health and well-being includes the ability to self-regulate emotionally, mentally, behaviorally and develop healthy relationships with peers and teachers. Better mood, coping with emotions and coping with stress are important for adolescents' development of life mastery skills and well-being. "Emotional regulation" as a method of communicating with emotions, as a well-known concept, refers to the way individuals manage an experience and express their emotions. In other words, emotional regulation describes the ability to both adapt emotional responses to socially accepted expressions and also allow flexibility in an individual's responses.

It has been stated that doing yoga can improve emotional regulation and the ability of individuals to give more adaptive responses. Miller et al. found that practicing yoga increases the ability to regulate emotional, cognitive, and somatic impulses and experiences. Similarly, in a review article on yoga and emotion regulation, Menezes et al. concluded: "Emerging evidence suggests that yoga may help promote healthier psychological responses, demonstrating its potential as an emotion regulation strategy". Other researchers have found that yoga in schools leads students to improve their mood and self-regulation skills and thus have better resilience. Yoga promotes awareness and acceptance and is a method for teaching young people to be more aware and aware of their own breath, body and mind. Studies have shown that yoga can reduce anxiety and improve emotion regulation skills among children and adolescents. Practicing yoga improves the mental health and well-being of teenagers and young adults, as well as increases their awareness of their bodies, minds, emotions, and response patterns. They suggest that "it occurs through interaction between activities that can lead to the development or enhancement of emotion regulation skills".

These authors found that attention regulation (via the prefrontal cortex), acceptance, regulation of autonomic activity (reduced anxiety and arousal), and endocrine responses underlie the relationship between yoga and emotion regulation. Increased awareness of themselves and their emotions can be valuable for teens to build resilience and improve their mental health and well-being.

Focusing on emotions is valuable because "how a person feels, reacts, and expresses emotions can have both short-term and long-term effects on physical and mental health" (13). This is explained by mechanisms such as reappraisal, attention regulation, self-monitoring, self-awareness, and regulation of the autonomic nervous system. Because yoga reduces negative emotions such as anxiety, anger, and depression, teens are likely to result in less conflict and stress in their lives. It is thought that it is also important for young people to accept difficult feelings and to be able to accept and approve these feelings. When negative emotions are acknowledged and witnessed, they often dissolve or transform, and the process allows the individual to learn about their limits, preferences, and needs. Processing emotions in this way allows a person to be honest with oneself and can contribute to healthier development. Therefore, yoga appears to be a useful well-being tool and practice that schools should adopt, as it can increase life skills for students such as concentration, memory, relational skills, and decision-making that are affected by emotions. Emotional well-being is important for learning in life and school. As noted earlier, research supports such a view, but more research is needed to understand how and why yoga should be offered to young people in their schools. However, it is suggested that researchers further explore the role of yoga in the management of emotions, both in terms of emotional processing and regulation of emotions. The role of yogic breathing (pranayama) as part of a holistic perspective on yoga, and specifically the role of yoga in the relationship between being with emotions, regulating emotions, and how it relates to change, should be further explored.

It has been described in the literature that care should be taken to avoid possible harm to individuals associated with the use of unhealthy weight control behaviors among young adults and women with obesity. Yoga's intent to strengthen and support a positive sense of self makes it a particularly viable strategy for healthy weight management for women and those at high risk for poor body image. Finally, it has been reported that reductions in perceived stress may mediate the effects of participation in a yoga program on negative emotional and behavioral problems. It has been suggested that future studies may also assess the extent to which exposure to stress and trauma may affect youth's participation in and benefit from mindfulness and yoga interventions.

Considering all the suggestions and research needs in the literature, this study was planned to examine the improvement in self-esteem, life satisfaction, body image, anxiety, depression and cognitive emotion regulation levels of university students after their participation in the yoga program provided to them in the school environment and to compare them with students who do not do yoga. In the study, it is planned to investigate the pre-exam anxiety levels of university youth who regularly practice yoga.

ELIGIBILITY:
Inclusion Criteria:

* students of Istanbul Medipol University,
* filling out all the scale questions
* agree to participate in the study

Exclusion Criteria:

* pregnancy
* having mental problems perceiving verbal commands
* having a concomitant disease that will hinder exercise and physical activity

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Emotion Regulation Questionnaire | up to 14 weeks
  Consisting of 36 items, the scale has nine subscales. Each subscale consists of four items. The five-point Likert-type scale is evaluated between 1 (never) and 5 (always). The score of each subscale varies between 4 and 20 and scoring is done accordingly. High scores obtained from the subscales indicate that the strategy determined by that subscale is used more.
The State-Trait Anxiety Inventory (STAI) | up to 14 weeks
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress. Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. The STAI is appropriate for those who have at least a sixth-grade reading level.
Body Cathexis Scale (BCS) | up to 14 weeks
  The form includes 40 items, each of which is related with an organ or a body zone (arm, leg, face, etc.) or with a function. Each item is rated between 1 and 5 points ("don't like at all," "don't like," "undecided," "like," and "like very much"), resulting in a total score between 40 and 200. The total score corresponds to the level of satisfaction with one's own body.
Satisfaction with Life Scale (SWLS) | up to 14 weeks
  Subjective well-being is conceptualised as consisting of two major components: the emotional or affective component and the judgment or cognitive component. The SWLS was designed to measure the judgment component. Scores consist of a raw score (between 5 and 35). Higher scores represent higher life satisfaction. Scorers can be assigned into six well-being categories and interpretative text in provided for each.
Rosenberg Self-Esteem Scale (RSES): | up to 14 weeks
  It consists of 10 items in total, 5 of which are positive expressions and 5 negative. Scores are given from "strongly disagree" (0) to "strongly agree" (3). A high total score demonstrated high self-esteem, a low score low self-esteem.
Test Anxiety Inventory | up to 14 weeks
  TAI was designed to measure anxiety in high school and university students. It consists of two subgroups: measurement of worry (TAI-W) and measurement of emotional distress (TAI-E). There are eight items in TAI-W, the inventory for measuring worry, eight items in TAI-E, the subscale focusing emotionality, and four items in TAI-T, a subscale for measuring total anxiety score. The respondents choose from the following options in Likert's four point scale: (1) almost never, (2) sometimes, (3) often, or (4) almost always. The values of the Cronbach Alpha coefficient of the original TAI were as follows: 0.96 for TAI-T, 0.91 for TAI-W, and 0.91 for TAI-E.
Three-factor Eating Questionnaire (TFEQ-R21) | up to 14 weeks
  The TFEQ-R21 (see Appendix) asks participants to respond to 21 questions on a four-point Likert scale for items 1-20 and on an eight-point numerical rating scale for item 21. Responses to each of the items are given a score between
  1 and 4. Before calculating domain scores, items 1-16 were reverse coded and item 21 was recoded as follows: 1-2 scores as 1; 3-4 as 2; 5-6 as 3; 7-8 as 4. Domain scores were then calculated as a mean of all items within each domain; hence, domain scores also ranged from 1 to 4 (CR (six items), UE (nine items) and EE (six items)), with higher scores being indicative of greater CR, UE and EE.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medipol University, Istanbul, Turkey (Türkiye)